CLINICAL TRIAL: NCT01355718
Title: A 26-week, Multicentre, Open-labelled, Non-randomised, Non-interventional, Observational, Safety Study of NovoNorm® (Repaglinide) and Insulin Analogue Combination Therapy in Type 2 Diabetes in Korea
Brief Title: Observational, Safety Study of NovoNorm® (Repaglinide) and Insulin Analogue Combination Therapy in Type 2 Diabetes in Korea
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-3905; U1111-1119-9152 (Other: WHO)
Record Dates: First submitted 2011-05-13; First posted 2011-05-18 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repaglinide
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — The dosage and frequency, as well as later changes to either dose, frequency or add-on medication (if applicable), will be determined by the physician, according to the patient's requirements.

SUMMARY:
This trial is conducted in Asia. The primary objective of this study is to evaluate the clinical safety profile during 26 weeks of NovoNorm® (repaglinide) and insulin analogue combination therapy in type 2 diabetes under normal clinical practice conditions in Korea while the secondary objective is to evaluate the safety and efficacy after 13 and 26 weeks of NovoNorm® and insulin analogue combination therapy in type 2 diabetes under normal clinical practice conditions in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol.)
* Patients with type 2 diabetes mellitus
* Patients who are currently treated with NovoNorm® alone or in combination with metformin or TZD
* Age: at least 18 years old
* Patients who will be prescribed with insulin analogue in addition to current NovoNorm® (with/without metformin/TZD) treatment at the discretion by the Physician

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Previous participation in this study. Participation is defined as screened
* Patients who have been treated with insulin preparations (including insulin analogues) previously
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Patients who are unlikely to comply with protocol requirements, e.g. uncooperative attitude, inability to return for the final visit
* Any other disease or condition that the Physician feels would interfere with study participation or evaluation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are currently treated with NovoNorm® alone or in combination with metformin or TZD (thiazolidinedione) and will be additionally prescribed with insulin analogue at the discretion of the physicians will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious Adverse Drug Reactions (SADRs) including major (serious) hypoglycaemic episodes | weeks 0-26

SECONDARY OUTCOMES:
Incidence of Adverse Drug Reactions (ADRs) | week 13 and 26
Incidence of Adverse Events (AEs) | week 13 and 26
Incidence of Serious Adverse Event (SAEs) | week 13 and 26
Change in HbA1c | after 13 and 26 weeks of NovoNorm® and insulin analogue combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com